CLINICAL TRIAL: NCT06590311
Title: Autonomic Modulation in Patients Undergoing Assisted Mechanical Ventilation: Comparison Between PAV+ and PSV
Status: Not yet recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Alessandri, Professor, University of Roma La Sapienza
Other Study IDs: RIA24.2
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mechanical Ventilation Weaning
Keywords: mechanical ventilation weaning; heart rate variability; autonomic modulation; PAV+

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PSV
  Interventions: Diagnostic Test: Heart Rate Variability
- PAV+
  Interventions: Diagnostic Test: Heart Rate Variability

INTERVENTIONS:
Diagnostic Test: Heart Rate Variability — Heart rate variability evaluation through different domains

SUMMARY:
The aim of the study is to investigate autonomic modulation in terms of heart rate variability (i.e., HRV) in patients undergoing assisted mechanical ventilation in PSV mode, compared to patients assisted in PAV+ mode. The hypothesis is that the greater patient-ventilator synchrony of the latter mode may represent an advantage in reducing the imbalance of autonomic modulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU, ≥18 years old, undergoing invasive controlled mechanical ventilation for at least 72 hours, eligible for assisted support but not yet ready for extubation or spontaneous breathing.

Exclusion Criteria:

* Successful completion of a spontaneous breathing trial (SBT) and spontaneous breathing within 24 hours of enrollment
* Acute ischemic heart disease, cardiac rhythm abnormalities, and/or patients with pacemakers and/or treated with anti-arrhythmic drugs
* Hemodynamic instability
* Chest drainage
* Severe anemia (Hb <7g/dL)
* Pregnancy
* Severe head trauma, dementia
* High spinal cord injury
* Neuromuscular disorders
* Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated ICU patients ready to be weaned
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
LF dominion | 30 min
  To evaluate the difference in the LF domain between patients assisted in PSV and those assisted in PAV+ at T1 (30 minutes).

SECONDARY OUTCOMES:
Other domains | 30 min to 72 hours
  To evaluate the difference in other HRV domains between patients assisted in PSV and those assisted in PAV+ at different time points.
Clinical outcomes | 28 days
  Correlation of HRV parameters with days of assisted ventilation and total ventilation, hospital length of stay (H-LOS) and ICU length of stay (ICU-LOS), mortality, organ dysfunction, delirium, supraventricular and ventricular arrhythmias, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico Umberto I, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided